CLINICAL TRIAL: NCT00969683
Title: Comparison Between Left Double-lumen Tube With or Without a Carinal Hook During Lung Surgery
Brief Title: Double-Lumen Tube With or Without a Carinal Hook
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/21
Record Dates: First submitted 2009-08-28; First posted 2009-09-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double lumen tube without a hook (Active Comparator): Broncho-Cath™, Mallinckrodt France, Parc d'Affaires Technopolis, 3 avenue du Canada, Bât Sigma, Les Ulis, 91975 Courtaboeuf Cedex
  Interventions: Device: Tracheal intubation
- Double lumen tube with a hook (Experimental): Broncho-Cath™, Mallinckrodt France, Parc d'Affaires Technopolis, 3 avenue du Canada, Bât Sigma, Les Ulis, 91975 Courtaboeuf Cedex
  Interventions: Device: Tracheal intubation

INTERVENTIONS:
Device: Tracheal intubation — Tracheal intubation using a Double lumen tube without a hook
  Arms: Double lumen tube without a hook
Device: Tracheal intubation — Tracheal intubation with a Double lumen tube with a hook
  Arms: Double lumen tube with a hook

SUMMARY:
Most teams use a left double-lumen tube. The double-lumen tube is available with or without a carinal hook. The hook is supposed to facilitate the positioning of the tube and avoid the mobilization of the tube during surgery. The use of double-lumen tubes with a hook is large in Europe and quite unknown in US. The literature is poor, containing only few case reports.

The purpose of this research is to compare the two types of left double-lumen tube.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for lung surgery requiring one-lung ventilation

Exclusion Criteria:

* pregnancy
* ASA class 4
* prevision of difficult intubation or of pulmonary aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
time required to initially position the assigned tube | end of anesthesia

SECONDARY OUTCOMES:
degree of lung collapse | end of anesthesia
number of intraoperatively FOB examinations | end of anesthesia
Glottic or tracheo-bronchial lesion | end of hospitalisation
Sore throat or hoarse voice | end of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Service d'Anesthésie, Hôpital Foch, Suresnes, France

REFERENCES:
- [Derived] Dumans-Nizard V, Parquin JF, Moyer JD, Dreyfus JF, Fischler M, Le Guen M. Left double-lumen tube with or without a carinal hook: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jun;32(6):418-24. doi: 10.1097/EJA.0000000000000201. PMID 25489763